CLINICAL TRIAL: NCT07272343
Title: A Study on the Impact of Semaglutide Compared to Energy Restriction on Type 2 Diabetes Combined With Metabolic-associated Fatty Liver Disease and Its Molecular Mechanisms
Brief Title: The Impact of Semaglutide Compared to Energy Restriction on Type 2 Diabetes
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Second Affiliated Hospital of Nanchang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022efyA04
Record Dates: First submitted 2025-11-16; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: Type 2 Diabetes Mellitus (T2DM); Semaglutide; Caloric Restriction
Keywords: Type 2 Diabetes Mellitus; semaglutide; Caloric Restriction
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — semaglutide; Caloric Restriction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- semaglutide group (Experimental): The semaglutide group received weekly subcutaneous semaglutide (0.25 mg for weeks 1-2, 0.5 mg for weeks 3-4, and 1.0 mg for weeks 5-12).
  Interventions: Drug: semaglutide
- caloric restriction group (Active Comparator): The caloric restriction group followed a gender-specific daily caloric restriction (1,500-1,800 kcal for males; 1,200-1,500 kcal for females).
  Interventions: Behavioral: caloric restriction

INTERVENTIONS:
Drug: semaglutide — The semaglutide group received weekly subcutaneous semaglutide (0.25 mg for weeks 1-2, 0.5 mg for weeks 3-4, and 1.0 mg for weeks 5-12).
  Arms: semaglutide group
Behavioral: caloric restriction — The caloric restriction group followed a gender-specific daily caloric restriction (1,500-1,800 kcal for males; 1,200-1,500 kcal for females).
  Arms: caloric restriction group

SUMMARY:
To evaluate the effects of subcutaneous injection of semaglutide for 12 weeks on patients with type 2 diabetes mellitus (T2DM), compared with concurrent energy-restricted management, on glycemic control, weight loss, inflammatory markers, liver fat content, and other parameters. The study also observed the subcutaneous and visceral fat of the participants and explored the molecular mechanisms of action, providing high-quality evidence-based support for the timing and targets of intervention in this population.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years;
2. BMI≥25 kg/m²;
3. Diagnosed as type 2 diabetes mellitus patients according to the "Guidelines for the Prevention and Treatment of Type 2 Diabetes in China (2020 Edition)";
4. HbA1c≤8.5%;
5. Duration of diabetes ≤3 months, and no use of antihyperglycemic drugs;
6. Willing to participate in this study, and after full informed consent, agrees to strictly follow the treatment plan and promises to attend follow-up visits on time, and signs the informed consent form.

Exclusion Criteria:

1. BMI < 25 kg/m²;
2. Age < 18 years, or > 75 years;
3. History of type 1 diabetes, acute pancreatitis, or diabetes secondary to pancreatectomy;
4. History of bariatric surgery or planned bariatric surgery, or currently attempting weight loss within the past 3 months, or use of weight-loss medications within the past 3 months;
5. Use of GLP-1 receptor agonists, sodium-glucose cotransporter 2 inhibitors, dipeptidyl peptidase-4 inhibitors, thiazolidinediones, or other related drugs within the past 3 months;
6. Pregnant or breastfeeding women, or those planning to conceive during the study period;
7. Patients with severe diseases of important organ systems, such as severe cardiovascular and cerebrovascular diseases, respiratory diseases, gastrointestinal diseases, renal insufficiency, hematologic diseases, neurological diseases, or malignancies;
8. Personal or family history of medullary thyroid carcinoma;
9. Patients with severe mental disorders or communication barriers that prevent accurate understanding of the study content and compliance with the trial procedures.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-02-10 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
HbA1c | From enrollment to the end of treatment at 12 weeks
  glycated hemoglobin
FPG | From enrollment to the end of treatment at 12 weeks
  fasting plasma glucose
2hPG | From enrollment to the end of treatment at 12 weeks
  2-hour postprandial glucose

SECONDARY OUTCOMES:
HOMA-IR | From enrollment to the end of treatment at 12 weeks
  homeostasis model assessment of insulin resistance
TC | From enrollment to the end of treatment at 12 weeks
  total cholesterol
TG | From enrollment to the end of treatment at 12 weeks
  triglycerides
LDL-C | From enrollment to the end of treatment at 12 weeks
  low-density lipoprotein
HDL-C | From enrollment to the end of treatment at 12 weeks
  high-density lipoprotein

CONTACTS AND LOCATIONS:
Locations (1):
- Minde road No.1, Jiangxi, Nanchang, China

IPD SHARING:
Plan to Share IPD: No
Some of the data involves patient privacy. If there is a need to share the data, please contact the relevant researchers of this project.